CLINICAL TRIAL: NCT07070297
Title: A Single-Arm Study to Evaluate the Effect on Airway Hyperresponsiveness, Safety, Immunogenicity, Pharmacokinetics, and Pharmacodynamics Characteristics of XKH001 Injection in Patients With Allergic Asthma
Brief Title: A Single-Arm Phase Ic Clinical Study of XKH001 Injection in Patients With Allergic Asthma After Multiple Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Kanova Biopharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XKH001-01-Ic
Record Dates: First submitted 2024-12-23; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Asthma Patients
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: The screening period will not be more than 28 days (i.e., 4 weeks). The treatment period will be 12 weeks, and the follow-up period will be 12 weeks.
  All recruited patients with allergic asthma will undergo various screening procedures within 28 days prior to the first dose, and those who pass the screening will be sequentially enrolled.
  Patients who are enrolled in the study will be admitted to the study site on the day before each scheduled dose (D-1, D28, and D56) to complete the necessary pre-dose safety assessments and receive XKH001 subcutaneous (SC) injections on D1, D29, and D57.
  The patient will undergo regular safety assessment procedures (AE/SAE, vital signs, physical examination, laboratory tests, 12-lead electrocardiogram (ECG), etc.), FeNO, pulmonary function tests (FEV1 PD20 Mch), sputum induction, and other blood sample collections (PK, PD, and ADA) during the treatment period (D1-D85) and the subsequent 12-week follow-up period (~D169).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experiment (Experimental): Patients who are enrolled in the study will be admitted to the study site on the day before each scheduled dose (D-1, D28, and D56) to complete the necessary pre-dose safety assessments and receive XKH001 subcutaneous (SC) injections on D1, D29, and D57.
  Interventions: Drug: XKH001 Injection

INTERVENTIONS:
Drug: XKH001 Injection — Dosage: 600 mg Q4W (D1, D29 and D57) Method of administration: the drug will be administered by SC injection in an area 3 cm away from and within 5 cm around the umbilicus of the abdomen. Sites with skin damage, inflammation, ulceration, rash and scar should be avoided. Subjects should be closely observed for reactions within 4 h after dosing.

SUMMARY:
This study is a single-arm, open-label clinical study. A total of 12 patients with allergic asthma are planned to be enrolled to receive XKH001 600 mg Q4W administration for the assessment of the safety, immunogenicity, PK, and PD characteristics of multiple doses.

DETAILED DESCRIPTION:
This study is a single-arm, open-label clinical study. A total of 12 patients with allergic asthma are planned to be enrolled to receive XKH001 600 mg Q4W administration for the assessment of the safety, immunogenicity, PK, and PD characteristics of multiple doses.

The screening period will not be more than 28 days (i.e., 4 weeks). The treatment period will be 12 weeks, and the follow-up period will be 12 weeks.

All recruited patients with allergic asthma will undergo various screening procedures within 28 days prior to the first dose, and those who pass the screening will be sequentially enrolled.

Patients who are enrolled in the study will be admitted to the study site on the day before each scheduled dose (D-1, D28, and D56) to complete the necessary pre-dose safety assessments and receive XKH001 subcutaneous (SC) injections on D1, D29, and D57.

The patient will undergo regular safety assessment procedures (AE/SAE, vital signs, physical examination, laboratory tests, 12-lead electrocardiogram (ECG), etc.), FeNO, pulmonary function tests (FEV1 PD20 Mch), sputum induction, and other blood sample collections (PK, PD, and ADA) during the treatment period (D1-D85) and the subsequent 12-week follow-up period (~D169).

Visits and procedures at screening, treatment, and follow-up are detailed in the Schedule of Assessment.

If a subject discontinues treatment prematurely, the "Early Withdrawal" visit and all procedures will be performed, the same as D169.

If asthmatic patients test positive for seasonal allergens (such as pollen), they should avoid the allergy season when enrolling in the study.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in the study, a subject must meet all of the following criteria:

  1. Subjects who voluntarily sign a written informed consent form (ICF) and are able to complete the study as required by the protocol;
  2. Male or female subjects aged 18 to 65 years (inclusive), with a body mass index (BMI) between 18 and 30 kg/m2 (inclusive);
  3. Subjects diagnosed with asthma according to the Guidelines for the Prevention and Treatment of Bronchial Asthma (China) 2020 with an asthma course (since the first incidence) of at least 6 months and meet the following requirements at the same time:

     Subjects with a positive reaction to at least 1 type of aeroallergen (such as dust mites, pollen, mold, or animal hair) in the skin prick test or allergen-specific IgE testing record before screening or during screening; Subjects with the upper limit of normal (ULN) at the site ≤ total serum IgE ≤ 1000 IU/mL at screening; Subjects with the bronchial provocation test FEV1 PD20 Mch ≤ 1.075 mg; Subjects with FEV1 ≥ 70% of the predicted value at screening;
  4. Subjects with occasional asthma symptoms (≤ 2 times/week), treated only with ICS-LABA inhalation (Symbicort®, budesonide and formoterol fumarate powder for inhalation, 1 inhalation per dose) as needed. The subject does not need to use other asthma medications on a daily basis, and other asthma medications have been discontinued before screening:

     Inhaled and nasal corticosteroids should be discontinued for 4 weeks; Leukotriene receptor antagonists should be discontinued for 2 weeks; Long-acting β-receptor agonists should be discontinued for 2 weeks; Anticholinergic drugs should be discontinued for 2 weeks; Antihistamines should be discontinued for 2 weeks; Theophylline drugs should be discontinued for 1 week.
  5. Subjects with normal laboratory test and 12-lead ECG results or with abnormalities determined by the investigator not to be clinically significant at screening;
  6. Women of childbearing potential must have a negative pregnancy test result and not be in the lactation period at screening; regardless of sex, all participants must agree to have no plans for reproduction during the study and within 6 months after the study, voluntarily adopt effective contraception measures, and have no plans for sperm/egg donation.

Exclusion Criteria:

* Subjects who meet any of the following criteria must be excluded from this study:

  1. Subjects who are current smokers or with a smoking history of > 10 pack-years. Subjects who have quit smoking need to have quit smoking for at least 12 months before enrollment;
  2. Subjects with hospitalization or emergency visits due to respiratory system and/or asthma-related conditions within 6 months before screening;
  3. Subjects with worsening or exacerbation of asthma, or the use of systemic glucocorticoid therapy within 6 weeks before or during screening;
  4. Subjects with a history of alcoholism or drug abuse;
  5. Subjects who are allergic to the investigational product or any component of the formulation of the investigational product or have a history of allergy to protein drugs;
  6. Subjects with elevated total IgE due to reasons other than allergens (e.g. parasitic infections and hematological disorders);
  7. Subjects who have undergone allergen-specific immunotherapy or used immunosuppressants within 3 months before screening;
  8. Subjects who have used biologics (such as monoclonal antibodies), including investigational biologics, within 6 months before screening;
  9. Subjects who have received any anti-IgE antibody treatment or bronchial thermoplasty within 12 months before screening;
  10. Subjects who have received live (attenuated) viral/bacterial vaccines or intravenous (IV) immunoglobulins (IgG) within 4 weeks before screening;
  11. Subjects with respiratory system infection or have received a major surgery within 8 weeks before screening;
  12. Subjects with a combination of other lung diseases such as COPD, bronchiectasis, or lung fibrosis;
  13. Subjects with a history of contraindications to choline, such as myocardial infarction or stroke within the past 3 months, known heart disease, uncontrolled hypertension, aortic or brain aneurysm;
  14. Subjects with neoplasm malignant within 5 years before screening or current neoplasm malignant;
  15. Subjects with a history of autoimmune diseases, known family history of inherited immunodeficiency disorders, or recurrent infections suggestive of possible immunodeficiency;
  16. Subjects who had or currently have active tuberculosis, or active infection requiring hospitalization or IV antibiotic treatment within 3 months before screening;
  17. Subjects with positive HBsAg in 5 items of hepatitis B serology (if HBsAg is negative, HBcAb is positive, and HBsAb is negative, HBV-DNA quantitative test is required to be performed [the subject will be excluded if the test result is positive]), hepatitis C antibody, treponema pallidum antibody, and HIV antigen/antibody;
  18. Subjects who have participated in other investigational drug clinical studies within 30 days or 5 half-lives of the study drug (whichever is longer). If a subject has received an investigational drug of a biological product, e.g., a monoclonal antibody, the subject is required to have received the biological product at least 6 months before the screening visit;
  19. Subjects with severe, progressive, or uncontrolled diseases such as liver, kidney, gastrointestinal, cardiovascular, hematopoietic, genitourinary, endocrine, nervous, immune system disorders, and other conditions that investigators consider unsuitable for inclusion in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma. | Day43, Day85
  Changes from baseline in FEV1 PD20 Mch after treatment
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.1 | Day169
  Incidence of AEs/SAEs
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.2 | Day169
  Severity of AEs/SAEs

SECONDARY OUTCOMES:
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.1 | Day169
  Incidence of ADAs and NAb [detect NAb when ADA positive];
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.2 | Day169
  FeNO (exhaled nitric oxide concentration);
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.3 | Day169
  Total IgE;
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.4 | Day169
  Levels of IL-25-related cytokines in sputum supernatants (same as serum).
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.6 | Day169
  Cmax,ss,
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.7 | Day169
  Cmin,ss
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.8 | Day169
  Cavg,ss
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.9 | Day169
  AUC0-inf,ss
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.10 | Day169
  AUC0-t,ss,
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.11 | Day169
  Tmax,ss,
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.12 | Day169
  t1/2,ss
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.13 | Day169
  AUCtau,
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.14 | Day169
  %AUCex
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.15 | Day169
  λz,ss
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.36 | Day169
  Vz,ss/F
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.16 | Day169
  CLss/F
To evaluate the effect on airway hyperresponsiveness and safety of multiple doses of XKH001 injection in patients with allergic asthma.17 | Day169
  MRT;
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.20 | Day169
  LYM ratios in sputum;
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.22 | Day169
  Whole blood EOS count
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.23 | Day169
  Whole blood NEU count
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.24 | Day169
  Whole blood LYM count
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.25 | Day169
  Whole blood MON count;
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.26 | Day169
  Levels of IL-25 in serum
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.27 | Day169
  Levels of TARC in serum
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.28 | Day169
  Levels of IL-8 in serum
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.29 | Day169
  Levels of MIP1β in serum
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.30 | Day169
  Levels of Eotaxin in serum
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.31 | Day169
  Levels of CXCL1 (KC/GROα) in serum
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.32 | Day169
  Levels of Eotaxin-3 in serum
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.33 | Day169
  Levels of IL-4 in serum
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.34 | Day169
  Levels of IL-5 in serum
To evaluate the immunogenicity, PK characteristics, and PD characteristics of multiple doses of XKH001 injection in patients with allergic asthma.35 | Day169
  Levels of IL-13 in serum;

CONTACTS AND LOCATIONS:
Overall Officials: Wen Li, Dr, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No